CLINICAL TRIAL: NCT01444885
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Therapeutic Exploratory Study to Evaluate the Efficacy and Safety of PletaalÒ(Cilostazol) in Subjects With Vasospastic Angina (STELLA)
Brief Title: Evaluate the Efficacy and Safety of Pletaal (Cilostazol) in Subjects With Vasospastic Angina
Acronym: STELLA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STELLA
Record Dates: First submitted 2011-09-27; First posted 2011-10-03 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Variant Angina
Keywords: Variant angina; Cilostazol
MeSH Terms: conditions — Angina Pectoris, Variant | interventions — Amlodipine; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cilostazol (Experimental): To investigate the efficacy and safety of Pletaal(Cilostazol) in comparison with placebo for 4 weeks in vasospastic angina patients who have an insufficient response to Amlodipine (Calcium channel blocker).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 2 weeks treatment of Cilostazol 100mg, or placebo oral tablets bid after 2 weeks treatment of Cilostazol 50mg, or placebo oral tablets bid (Total 4 weeks)
  Other Names: Amlodipine; Nitroglycerin

SUMMARY:
The objective of this study is to investigate the efficacy and safety of Pletaal (Cilostazol) in comparison with placebo for 4 weeks in vasospastic angina patients who have an insufficient response to Amlodipine (Calcium channel blocker).

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-Blind, Placebo-controlled, Parallel group, Therapeutic exploratory Study.

The subject who has at least an episode of chest pain weekly despite Amlodipine 5mg once a day (qd) taking during 2 weeks will have treatment of Pletaal (Cilostazol) or Placebo for 4 weeks. Pletaal (Cilostazol) is taken 100mg oral tablets two times a day (bid) during 2 weeks after dosing of Pletaal (Cilostazol) 50mg oral tablets bid during 2 weeks. Placebo of Pletaal (Cilostazol) is used as the control medication.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over the age of 20 and under the age of 80
2. Diagnosis of vasospastic angina
3. At least one episode of chest pain weekly during the Amlodipine run in period for 2 weeks

Exclusion Criteria:

1. Currently taking or has taken Cilostazol within the last 3 month before the screening.
2. Taking oral antiplatelet agents such as Aspirin, Clopidogrel after Amlodipine run-in period.
3. Oral anticoagulants such as Warfarin within the last a month before the screening.
4. Currently taking any of the following medications or has taken any of the following medications within the last a week before the screening:

   * Other Calcium channel blockers than Amlodipine
   * Beta-blocker, or Alpha-blocker
   * Oral Nitrate, Nicorandil, except sublingual Nitroglycerin as required(PRN)
   * Vitamin E preparations
   * Estrogens
5. History of Myocardial infarction or Myocardial infarction by vasospastic angina at screening
6. History of life threatening vasospastic events such as ventricular tachycardia , ventricular fibrillation, or syncope
7. History of stroke, intracranial hemorrhage, or Transient Ischemic Attack(TIA)
8. Hemorrhage (hemophilia, capillary fragility, intracranial hemorrhage, upper gastrointestinal hemorrhage, urinary hemorrhage, hemoptysis, vitreous hemorrhage, etc.) or such tendency (active peptic ulcer, hemorrhagic stroke within past 6 months, a case hemorrhage is suspected by wound for surgery within 3 months, proliferative diabetic retinopathy and uncontrolled hypertension)
9. History of clinically significant hypersensitivity to the substances of Cilostazol, Amlodipine, Nitroglycerin or dihydropyridine
10. Patients with severe aortic valvular stenosis
11. History of shock
12. Hypotension of diastolic pressure < 90 mmHg at screening
13. History of clinically significant hypersensitivity to the substances of Nitrates
14. Patients with severe anemia of Hemoglobin ≤ 6.5 g/dl at screening
15. History of glaucoma
16. Electrocardiogram(ECG) abnormality precluding interpretation of ST change at screening
17. Congestive heart failure with less than 40% of left ventricular ejection fraction within the last 3 month before the screening or screening period
18. Atrial fibrillation or valvular heart disease, more than moderate severity
19. Suspected or identified spasm of left main coronary artery, result of coronary angiography or coronary angiography in the ergonovine induced coronary spasm provocation test
20. History of Coronary artery bypass graft(CABG) or percutaneous coronary intervention(PCI)
21. Tachycardia; Heart rate > 100 bpm, at Screening
22. Uncontrolled hypertension, defined as ≥ 160 mmHg systolic or ≥ 100 mmHg diastolic at Screening
23. Creatinine ≥ 1.5 mg/dL at screening
24. Aspartate transaminase (AST) or alanine transaminase (ALT) > 3 times the upper limit of normal (ULN) at screening
25. Platelet < 100,000 mm3 at screening
26. QT prolongation defined as baseline QTc > 450 msec for males or > 470 msec for females at Screening.
27. Women who have the possible of pregnancy, or positive urine or blood pregnancy test at screening
28. Women who are not using a reliable method of birth control, who are pregnant, or who are breast-feeding
29. Drug compliance of Amlodipine < 80% during the Amlodipine run in period for 2 weeks
30. Otherwise judged by the investigator to be inappropriate for inclusion in the trial.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Percent change of the chest pain frequency | A week before IP dosing and the final a week after IP dosing (average 6weeks)
  Collect the chest pain frequency data related with vasospastic angina episodes by subject diaries.
  Descriptive statistics (N, mean, standard deviation, minimum, median and maximum) will be presented by treatment group. ANCOVA will be performed between the treatment groups using the baseline (a week before IP dosing) as covariate.

SECONDARY OUTCOMES:
The chest pain frequency, the pain intensity, nitroglycerin consumption of the final a week after IP dosing from a week before IP dosing | A week before IP dosing and the final a week after IP dosing (average 6weeks)
  Descriptive statistics (N, mean, standard deviation, minimum, median and maximum) will be presented by treatment group. ANCOVA will be performed between the treatment groups using the baseline (a week before IP dosing) as covariate. The subject who has no chest pain will be regarded as the total pain intensity and the average pain intensity are '0'. The subject who has taken no nitroglycerin will be regarded as taking '0' tablet.

CONTACTS AND LOCATIONS:
Overall Officials: June Hong Kim, MD, Principal Investigator — Pusan National University Yansan Hospital
Locations (10):
- South Korea (10):
  - Keimyung University Dongsan Medical Center, Daegu
  - ChungNam Univ. Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Gyongsang National University Hospital, Jinjoo
  - Dong-A University Hospital, Pusan
  - Pusan National University Yansan Hospital, Pusan
  - Asan Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Shin ES, Lee JH, Yoo SY, Park Y, Hong YJ, Kim MH, Lee JY, Nam CW, Tahk SJ, Kim JS, Jeong YH, Lee CW, Shin HK, Kim JH. A randomised, multicentre, double blind, placebo controlled trial to evaluate the efficacy and safety of cilostazol in patients with vasospastic angina. Heart. 2014 Oct;100(19):1531-6. doi: 10.1136/heartjnl-2014-305986. Epub 2014 Jun 16. PMID 24934484